CLINICAL TRIAL: NCT03469232
Title: Effectiveness and Clinical Mechanism of Huanglian-Jiedu Decoction in Patients With Intense-exuberant Stomach Fire Syndrome (Acute Pericoronitis, Minor Recurrent Aphthous Stomatitis and Recurrent Herpes Simplex Labialis)
Brief Title: Effectiveness and Clinical Mechanism of Huanglian-Jiedu Decoction in Patients With Intense-exuberant Stomach Fire Syndrome
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhong Wang, Chief, China Academy of Chinese Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLJD-V3
Record Dates: First submitted 2018-02-28; First posted 2018-03-19 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Intense-exuberant Stomach Fire Syndrom; Acute Pericoronitis; Recurrent Aphthous Stomatitis; Recurrent Herpes Simplex Labialis
MeSH Terms: conditions — Stomatitis, Aphthous; Herpes Labialis | interventions — huanglian-jie-du decoction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Huanglian-Jiedu Decoction in acute pericoronitis (Experimental): All eligible patients entering this group will receive Huanglian-Jiedu Decoction(prepared as granule). 1 bag per time and twice a day for 5 days.
  Interventions: Drug: Huanglian-Jiedu Decoction
- Huanglian-Jiedu Decoction in recurrent aphthous stomatitis (Experimental): All eligible patients entering this group will receive Huanglian-Jiedu Decoction(prepared as granule). 1 bag per time and twice a day for 5 days.
  Interventions: Drug: Huanglian-Jiedu Decoction
- Huanglian-Jiedu Decoction in recurrent herpes simplex labialis (Experimental): All eligible patients entering this group will receive Huanglian-Jiedu Decoction(prepared as granule). 1 bag per time and twice a day for 5 days.
  Interventions: Drug: Huanglian-Jiedu Decoction

INTERVENTIONS:
Drug: Huanglian-Jiedu Decoction — Huanglian-Jiedu Decoction includes 4 kinds of Chinese herbs as following: Huanglian (Rhizoma Coptidis), Huangbo (Cortex Phellodendri), Huangqin (Scutellaria baicalensis) and Zhizi (Scutellaria baicalensis). All of them were prepared as granule.

SUMMARY:
This clinical research focus on evaluating the effectiveness of Huanglian-Jiedu Decoction in patients with intense-exuberant stomach fire syndrome (one of the common TCM syndrome)of acute pericoronitis,minor recurrent aphthous stomatitis and recurrent herpes simplex labialis,meanwhile, exploring the pharmacological mechanism and potential biomarkers of this traditional formula.

DETAILED DESCRIPTION:
Huanglian-Jiedu Decoction, as a traditional Chinese medicine formula，includes 4 kinds of Chinese herbs as following: Huanglian (Rhizoma Coptidis), Huangbo (Cortex Phellodendri), Huangqin (Scutellaria baicalensis) and Zhizi (Scutellaria baicalensis). Huanglian-Jiedu Decoction has been recorded to be effective in many diseases that belong to the syndrome of intense-exuberant stomach fire from thousands years of clinical practice, just like acute pericoronitis, minor recurrent aphthous stomatitis and recurrent herpes simplex labialis,etc. While its clinical pharmacological mechanism has not been clearly illustrated. In this study, the investigators focus on evaluating the effectiveness of Huanglian-Jiedu Decoction in patients with intense-exuberant stomach fire syndrome (including three disease: acute pericoronitis, minor recurrent aphthous stomatitis and recurrent herpes simplex labialis), and exploring the pharmacological mechanism and potential biomarkers of this traditional formula.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  1. Female or male patients.
  2. Age: 18 - 60 years.
  3. Meeting the diagnostic criteria of Intense-Exuberant Stomach Fire Syndrome according to the traditional Chinese medicine.
  4. Patient is willing to participate voluntarily and to sign a written patient informed consent.
* Disease-specific inclusion criteria for patients with acute pericoronitis:

  1. Patients with clinical diagnosis of acute pericoronitis and without treatment before the study began.
* Disease-specific inclusion criteria for patients with minor recurrent aphthous stomatitis:

  1. Patients with clinical diagnosis of minor recurrent aphthous stomatitis(MiRAS).
  2. A history of MiRAS for more than 6 months and an expectation that the ulcers normally take 5 or more days to resolve without treatment.
  3. Ulcer occurred less than 48h hours' duration without treatment.
* Disease-specific inclusion criteria for recurrent herpes simplex labialis

  1. Patients with clinical diagnosis of recurrent herpes simplex labialis.
  2. History of recurrent herpes labialis averaging 1 or more episodes per year.
  3. Onset of prodrome, erythema or vesicle within 48 hours without treatment.

Exclusion Criteria:

* General exclusion criteria:

  1. Patients with severe cardiac dysfunction on the grade of heart function over Ⅲ grade and/or liver function impairment with the value of ALT over 1.5-fold of normal value and/or renal dysfunction with the value over 133μmol/L.
  2. Patients who have serious, unstable, or clinically significant medical or psychological conditions, which, in the opinion of the investigator(s), would compromise the subject's participation in the study (including but not limited to arrhythmia, uncontrolled hypertension, diabetes, hepatitis, kidney failure, AIDS, cancer, etc.
  3. Women during pregnancy, lactation , breastfeeding or having child bearing potential without use an adequate method of birth control.
  4. Patients who known allergy to the study drug or the Huanglian (Rhizoma Coptidis), Huangbo (Cortex Phellodendri), Huangqin (Scutellaria baicalensis) and Zhizi (Scutellaria baicalensis ( Patients who are insufficiency of the spleen-yang according to the TCM should be exclude ).
  5. Patients participating in or having participated in other clinical studies in the 3 months prior to this clinical trial.
  6. Patients who are considered unreliable as to medication compliance or adherence to scheduled appointments.
* Disease-specific exclusion criteria for acute pericoronitis:

  1. Patients who smoked at least 20 cigarettes per day（heavy smokers）.
  2. Patients with fascial space infection of maxillofacial region or/and chronic periodontitis.
  3. Patients with periodontal disease in the region of the acute pericoronitis.
  4. Patients who had systemic administration of antibiotics within the past 4 weeks
* Disease-specific exclusion criteria for minor recurrent aphthous stomatitis(MiRAS):

  1. Patients with history of drug abuse within the past 6 months.
  2. Patients who smoked at least 20 cigarettes per day（heavy smokers）.
  3. Patients with ulcers as a manifestation of a systemic disease process such as ulcerative colitis, Behcet's syndrome, Reiter' s syndrome or immune deficiency.
  4. Patients who had systemic administration of antibiotics within the past 4 weeks or/ and had treatment with systemic steroid or immunomodulatory within 3 month before the study entry.
  5. Patients who had orthodontic braces or retainer that might contact with the ulcer.
* Disease-specific exclusion criteria for recurrent herpes simplex labialis:

  1. Patients with fever > 38.5℃, and / or blood WBC>11.0x109/L, and / or neutrophil >85%.
  2. Patients who had systemic administration of antibiotics within the past 4 weeks or/ and had treatment with immunomodulatory within 3 month before the study entry.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Intense-Exuberant Stomach Fire Syndrome scores | Day 0,Day 3,Day 5
  Intense-Exuberant Stomach Fire Syndrome scores were questionnaires that consists of basic symptoms and disease-specific symptoms that described in traditional Chinese medicine. The basic symptoms included feverish sensation, thirst that preferring cold drink, bad breath, flushed face, bound stool, scanty yellowish urine, red tongue with dry and yellowish fur, and the forceful or rapid pulse. The disease-specific symptoms included tooth or/and gums for acute pericoronitis, ulcer for recurrent aphthous stomatitis and herpes for recurrent herpes simplex labialis. Each symptom was assessed by the Visual Analogue Scale（VAS），where a higher score meant higher severity.

SECONDARY OUTCOMES:
Change from baseline of each symptom in Intense-Exuberant Stomach Fire Syndrome scores | Day 0,Day 3,Day 5
The proportion of patients whose Intense-Exuberant Stomach Fire Syndrome were disappeared | Day 0,Day 5
  The definition of "disappeared" is the scores of all the symptoms in Intense-Exuberant Stomach Fire Syndrome were 0 or the reduction in rate of Intense-Exuberant Stomach Fire Syndrome scores more than 90%
The proportion of patients who gain 50% reduction of Intense-Exuberant Stomach Fire Syndrome scores | Day 0,Day 5
  Reduction in rate of Intense-Exuberant Stomach Fire Syndrome scores =（The score of Intense-Exuberant Stomach Fire Syndrome before treatment - the score of Intense-Exuberant Stomach Fire Syndrome after treatment）/ The score of Intense-Exuberant Stomach Fire Syndrome before treatment×100%.
Change from baseline on toothache based on visual analogue scale(VAS)for acute pericoronitis | Day 0,Day 1,Day 2,Day 3,Day 4,Day 5
  Patients were asked to record the VAS each morning for 5 consecutive days prior to taking their medication.
Change from baseline on maximum mouth opening (MMO) for acute pericoronitis | Day 0,Day 3,Day 5
  To measure the amount of MMO, the inter-incisal distance between maxillary and mandibular right central incisors was recorded using a caliper.
Number of patients with trismu for acute pericoronitis | Day 0,Day 3,Day 5
  Patients were recorded to have trismus if the MMO was less than 40 mm.
Change from baseline on OHIP-14 measures for acute pericoronitis | Day 0,Day 3,Day 5
  Using the OHIP measures, the patients were asked to rate the impact of their oral health on 14 key areas of OHRQoL: "What effects do your teeth, gums, and/or mouth have on each of the 14 key areas of life quality (i.e., your comfort, your speech)?" These 14 items were subdivided into seven domains (subscales): functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability, and handicap. For the OHIP-14, the response categories were recorded on a five-point Likert scale: 0, never; 1, hardly ever; 2, occasionally; 3, fairly often; 4, very often. Higher scores in the OHIP-14 questionnaire indicated a poorer OHQoL.
Change from baseline of VAS on the pain of ulcer for minor recurrent aphthous stomatitis | Day 0,Day 1,Day 2,Day 3,Day 4,Day 5
  Patients were asked to record the VAS each morning for 5 consecutive days prior to taking their medication.
The proportion of patients with ulcer healing for minor recurrent aphthous stomatitis | Day 0,Day 3,Day 5
The sizes of ulcer for minor recurrent aphthous stomatitis | Day 0,Day 3,Day 5
  The investigators chose one of the largest ulcer and measured the maximum diameters and its vertical using a calibrated dental probe with millimeter markings. The two measurements were then multiplied to represent the size of the ulcer.
The number of days that the lesion was present (until loss of crust)for recurrent herpes simplex labialis | From the date of lesion or premonitory symptom present until the date of crust lose, which up to 28 days.
The proportion of patients with lesion healing for recurrent herpes simplex labialis | Day 3,Day 5
Change from baseline of VAS on the pain of lesions for recurrent herpes simplex labialis | Day 0,Day 1,Day 2,Day 3,Day 4,Day 5
  Patients were asked to record the VAS each morning for 5 consecutive days prior to taking their medication.

OTHER OUTCOMES:
High-sensitivity C-reactive protein（hs-CRP） | Day 0,Day 5
Evaluation of inflammatory cytokines | Day 0,Day 5
  The evaluation of inflammatory cytokines include IL-1α, IL-1β, IL-4, IL-6, IL-8, IL-10, IL-13, MIP-2, MCP-1, IFNγand TNF-α
Activity of sirtuins (SIRTs) | Day 0,Day 5
  Detection by qRT-PCR
GSH/GSSG ratios in plasma | Day 0,Day 5
Evaluation of oxidative stress parameters：SOD | Day 0,Day 5
Evaluation of oxidative stress parameters：MDA | Day 0,Day 5
Pyruvate Acid / Uric Acid ratios in plasma | Day 0,Day 5
Mass Spectrometry analyses for urine sample | Day 0,Day 5
  Mass Spectrometry analyses for urine sample include hypoxanthine, 1.7 - diphosphate sedoheptose, -5- riboflavin phosphate, urobilin, D - Ribose, ubiquinone, urinary lactate / pyruvate urine
Proteomic analyses for blood sample | Day 0,Day 5
Proteomic analyses for urine sample | Day 0,Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences
Locations (3):
- China (3):
  - Third affiliated hospital of Beijing University of traditional Chinese medicine, Beijing, Beijing Municipality
  - Dongfang Hospital Affiliated to Beijing University of traditional Chinese medicine, Beijing, Beijing Municipality
  - Affiliated Hospital to Chengdu University of traditional Chinese medicine, Chengdu, Sichuan